CLINICAL TRIAL: NCT02350218
Title: Open-label, Single Center, Randomized Clinical Trial to Evaluate Safety, Efficacy of Eglandin® (Alprostadil) 360㎍, 720㎍ in Living Donor Liver Transplanted Patient
Brief Title: Safety, Efficacy of Eglandin® in Living Donor Liver Transplanted Patient (PROVISION)
Acronym: PROVISION
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Giwon Song, Professor, Asan Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LSI-2014-0624
Record Dates: First submitted 2015-01-20; First posted 2015-01-29 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Evidence of Liver Transplantation
Keywords: Transplantation; Living donor; Eglandin; Alprostadil
MeSH Terms: interventions — Alprostadil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eglandin 720㎍ (Experimental): Eglandin® (Alprostadil) 720㎍
  Interventions: Drug: Eglandin
- Eglandin 360㎍ (Active Comparator): Eglandin® (Alprostadil) 360㎍
  Interventions: Drug: Eglandin

INTERVENTIONS:
Drug: Eglandin — Inject Eglandin 360㎍ or 720㎍ for 14 days in living donor liver transplanted patient
  Other Names: Alprostadil

SUMMARY:
The purpose of this study is to evaluate superiority of Eglandin® (Alprostadil) 720㎍compared to 360㎍ in terms of safety, efficacy in living donor liver transplant patient, peak AST levels followed by Eglandin administration were assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Primary living donor liver transplantation
2. Patient received modified right lobe graft
3. Aged between 19 to 65 years
4. Informed consent

Exclusion Criteria:

1. ABO incompatibility
2. Dual liver transplant patient from 2 donors
3. History of liver transplantation or other organ transplantation
4. Transplantation of other organ(s) at the time of liver transplantation
5. Use of artificial liver device prior to liver transplantation
6. UNOS status Ⅰor ⅡA
7. History of malignant tumor within 5 years
8. Not included in Milan liver transplant criteria for hepatocellular carcinoma
9. Patient with WBC < 2,000/mm3 or ANC < 900/mm3 or platelet < 30,000/mm3 at the time of screening
10. Patient exposed to severe systemic infection requiring treatment
11. Positive response for HIV in either donor or recipient
12. Prior administration of other investigational product within 30 days (or 5 times the half life) from date of screening
13. Women of childbearing age without effective contraception, breast feeding and pregnant women
14. Substance abuser, patient with metal disorder, and otherwise legally not eligible patient
15. Not eligible to participate at discrete of study investigator

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2015-03; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Peak AST level within 7 days of Eglandin administration | 7 days

SECONDARY OUTCOMES:
Area Under the Curve (AUC) of serum AST level within 5 days of Eglandin administration | 5 days
Absolute and relative (percent) change in peak AST level within 7 days of Eglandin administration from baseline | 7 days
Peak ALT levels within 7 days of Eglandin administration | 7 days
Change in blood flow rate of hepatic artery/vein/portal from baseline at 7th, 14th, 60th, and 120th day from first dose of Eglandin administration | 7th, 14th, 60th, and 120th day from first dose of Eglandin administration
Change in total bilirubin/AST/ALT from baseline at 7th, 14th, 30th, and 60th day from first dose of Eglandin administration | 7th, 14th, 30th, and 60th day from first dose of Eglandin administration
Peak total bilirubin levels within 7, 14, 30 and 60 days from first dose of Eglandin administration | 7, 14, 30 and 60 days from first dose of Eglandin administration
Time to total bilirubin recovery (within reference range) | day 2~14, day 30, 60,90, 120,150,180 from first dose of Eglandin administration
Transplant liver survival rate on Day 180 | Day 180
Incidence of hepatic artery/vein/portal thrombosis on Day 180 | Day 180
Safety (other laboratory test, vital sign, adverse event) evaluation | All visit(Screening, baseline, day 2~14, day 30, 60,90, 120,150,180)

CONTACTS AND LOCATIONS:
Overall Officials: Giwon Song, Professor, Principal Investigator — Asan Medical Center
Locations (1):
- Korea, Republic of, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No